CLINICAL TRIAL: NCT01504672
Title: A Randomized Controlled Pharmacist Intervention Study to Reduce Drug-related Problems and Readmissions Among Old People With Dementia
Brief Title: An Intervention Study to Reduce Drug-related Problems and Readmissions Among Old People With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Hugo Lovheim, Principal Investigator, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UmU-2011-148-31M
Record Dates: First submitted 2012-01-03; First posted 2012-01-05 (Estimated); Results first posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-10

CONDITIONS: Cognitive Impairment
Keywords: Drug related problems
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Medication Review

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Medication review (Experimental)
  Interventions: Other: Medication review
- Usual care (No Intervention)

INTERVENTIONS:
Other: Medication review — In the intervention, the pharmacist will evaluate:
  * Is there an indication for the drug?
  * Has the drug desired effect?
  * Is the dose correct and dosing scheme correct?
  * Side effects, contraindications, inappropriate drugs
  * Interactions
  * Treatment time
  * Cost effectiveness
  * Adherence to recommendation list
  * Problems with handling the drugs (for example crushing of the tablets)
  * Untreated indication
  * Double medications
  * Administration of drugs
  Arms: Medication review

SUMMARY:
The aim of this randomized controlled study is to investigate if medication reviews performed by a clinical pharmacist as part of a ward team can reduce drug related problems and reduce readmissions to hospital among elderly patients (≥65 years) with dementia and cognitive failure.

Four hundred and sixty patients will be recruited and randomized to control (usual care) and intervention group (enhanced service in which a pharmacist is part of the health care team).

Six months after the last patient of the 460 has been discharged the study will be closed. Data about the number of readmissions and visits to the emergency room will be collected during the six-month follow-up and also, the costs associated with each visit or admission. Time until institutionalization will be compared between intervention group and control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with dementia or cognitive impairment
* Patients ≥ 65 years

Exclusion Criteria:

* Patients previously admitted to the study wards during the study period

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 460 (Actual)
Dates: Start 2012-01; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Lövheim, MD, PhD, Principal Investigator — Umeå University, Umeå, Sweden
Locations (2):
- Sweden (2):
  - County hospital of Skellefteå, Skellefteå
  - Umeå University Hospital, Umeå

REFERENCES:
- [Derived] Gustafsson M, Sjolander M, Pfister B, Jonsson J, Schneede J, Lovheim H. Pharmacist participation in hospital ward teams and hospital readmission rates among people with dementia: a randomized controlled trial. Eur J Clin Pharmacol. 2017 Jul;73(7):827-835. doi: 10.1007/s00228-017-2249-8. Epub 2017 Apr 8. PMID 28391409

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group: Medication review: In the intervention, the pharmacist will evaluate:
  * Is there an indication for the drug?
  * Has the drug desired effect?
  * Is the dose correct and dosing scheme correct?
  * Side effects, contraindications, inappropriate drugs
  * Interactions
  * Treatment time
  * Cost effectiveness
  * Adherence to recommendation list
  * Problems with handling the drugs (for example crushing of the tablets)
  * Untreated indication
  * Double medications
  * Administration of drugs
- Control Group: Usual Care where no medication review is performed by clinical pharmacists
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 230 | 230
Completed | 212 | 217
Not Completed | 18 | 13

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group: An intervention as described is performed for the people in the intervention group.
- Control Group: No intervention is performed.
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 212 | 217 | 429
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 212 | 217 | 429
Age, Continuous [Mean (Standard Deviation); unit: years] | 83.1 (6.6) | 83.1 (6.6) | 83.1 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 133 | 138 | 271
  Male | 79 | 79 | 158
Region of Enrollment [Number; unit: participants]
  Sweden | 212 | 217 | 429
Medical history [Number; unit: participants]
  Heart failure | 72 | 54 | 126
  Hypertension | 116 | 105 | 221
  Cardiac arrhythmia | 62 | 58 | 120
  Diabetes Mellitus | 61 | 47 | 108
  COPD | 16 | 18 | 34
  Malignant disease, past or present | 27 | 20 | 47
  Myocardial infarction | 36 | 25 | 61
  Stroke, past | 50 | 46 | 96

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Readmitted Because of Drug Related Reasons
Time Frame: Six months follow-up
Measure: Number; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 212 | 217
Participants | 40 | 50

2. Secondary Outcome: Cost for Visits for Readmissions and to the Emergency Department Compared Between Patients in the Control Group and Intervention Group.
Description: To evaluate the economic impact of clinical pharmacist engagement in hospital ward teams for medication therapy management in older patients with dementia or cognitive impairments.
Time Frame: Six months follow-up
Measure: Mean (Standard Deviation); unit: Euro
Arm/Group | Medication Review | Usual Care
Number analyzed (Participants) | 212 | 217
Euro | 2340 (0) | 2630 (0)

3. Secondary Outcome: Number of Participants Institutionalized After Discharge, in Control Group and Intervention Group.
Time Frame: Six months follow-up
Population: Of the 460 people included in this study, 31 deceased before discharge. Of the remaining 429 persons, 146+158=304 persons lived at home, and these were included in the analysis. The remaining 125 were already living in nursing homes and were not included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 146 | 158
Participants | 17 | 24

4. Secondary Outcome: Frequency of Emergency Department Visits During the 6-month Follow-up.
Time Frame: Six months follow-up
Measure: Number; unit: All-cause emergency department visits
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 212 | 217
All-cause emergency department visits | 190 | 184

5. Secondary Outcome: Change in the Number of Participants With Potentially Inappropriate Medications, According to the Swedish National Board of Health and Welfare, at Admission and Discharge Between Intervention and Control Group
Description: Six drug-specific quality indicators as defined by the Swedish National Board of Health and Welfare were used to define use of Potentially inappropriate medications (PIMs) in this study. Four out of the six selected indicators belong to a group where drug-use should be as low as possible regardless of indication: anticholinergic drugs (as defined by the Swedish National Board of Health and Welfare, propiomazine, tramadol, and long-acting benzodiazepines. The two remaining indicators are classified as preparations for which correct and current indication is of particular importance: antipsychotic drugs (N05A except lithium) and Nonsteroidal Anti-Inflammatory Drugs (NSAIDs). In the present study, a PIM was defined as exposure to at least one of the drugs mentioned among the six quality indicators.
Time Frame: Index admission (at randomization) and index discharge (duration of index admission, mean days 8.7)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 212 | 217
Participants | 13 | 5

6. Post Hoc Outcome: Time From Discharge to Drug-related Readmission
Description: Time from discharge to drug-related readmission among the whole sample, post-hoc
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Medication Review | Usual Care
Number analyzed (Participants) | 212 | 217
days | 29.1 (0.30) | 28.1 (0.43)

ADVERSE EVENTS:
Arm/Group | Intervention Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/212 | 0/217
Other Adverse Events (participants affected / at risk) | 0/212 | 0/217

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No